CLINICAL TRIAL: NCT06574399
Title: Identification and Validation of Clinical Phenotypes in Staphylococcus Aureus Bacteremia and Their Association With Mortality and Development of Complicated Bacteremia
Acronym: FEN-AUREUS
Status: Recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-FENAUREUS-2022-01
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Staphylococcus Aureus Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine retrospectively whether different patient clinical phenotypes (adults and children) develop Staphylococcus aureus bacteremia.The main questions it aims to answer qre:

1. Evaluate its reproducibility and correlation with mortality
2. Derive and validate a simplified probabilistic model for phenotype assignment
3. External validation of the simplified probabilistic phenotype assignment model found and its association with mortality and development of complicated bacteremia in a prospective cohort
4. Apply microbiological, biochemical and immunological techniques to explain the physiopathological and genetic mechanisms underlying the phenotypes.

ELIGIBILITY:
FOR STANDARD STUDY:

Inclusion Criteria:

* Adults and children with clinically significant Staphylococcus aureus bacteremia (at least two classic systemic inflammatory response criteria: fever, tachycardia, tachypnea, lowered awareness, low blood pressure, leucocytosis/leucopenia, organ failure)

Exclusion Criteria:

* Patients with non-clinically significant bacteremia.
* Death within 48 hours after detection of bacteremia for the inclusion of retrospective cases, life expectancy less than 48 hours for the inclusion of retrospective cases, life expectancy less than 48 hours for the inclusion of retrospective cases.
* Patients under palliative sedation at the time of bacteremia report.
* Polymicrobial bacteremia.

FOR EXTENDED STUDY:

Inclusion Criteria:

* Adults with clinically significant Staphylococcus aureus bacteremia included in the Standard Study
* Selected at random as one of the model phenotypes until completing recruitment (only HUVM and HUVV)

Exclusion Criteria:

* Patients with non-clinically significant bacteremia.
* Death within 48 hours after detection of bacteremia for the inclusion of retrospective cases, life expectancy less than 48 hours for the inclusion of retrospective cases, life expectancy less than 48 hours for the inclusion of retrospective cases.
* Patients under palliative sedation at the time of bacteremia report.
* Polymicrobial bacteremia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with clinically significant Staphylococcus aureus bacteremia
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Determine whether different patient clinical phenotypes develop S. aureus bacteremia, evaluate its reproducibility and correlation with mortality and derive and validate a simplified probabilistic model for phenotype assignment | 1 month
  Analyze the ISAC (International Staphylococcus aureus collaboration) cohort from an international study (11 hospitals in five countries) on Staphylococcus aureus bacteremia (2590 cases)

SECONDARY OUTCOMES:
External validation of the simplified probabilistic phenotype assignment model found and its association with mortality and development of complicated bacteremia in a prospective cohort | 34 months
  Perform a multicenter prospective cohort study (Standard study): All patients who develop S. aureus bacteremia will be assigned a phenotype and followed up for six months to evaluate the differences in mortality and development of complicated bacteremia between phenotypes.
Apply microbiological, biochemical and immunological techniques to explain the physiopathological and genetic mechanisms underlying the phenotypes | 34 months
  Study the genetic (microorganism and patient), immunological, biochemical and microbiological variables in patients representative of the phenotypes selected in the prospective cohort in two hospitals (Extended Study)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: No